CLINICAL TRIAL: NCT01385384
Title: Evaluation of the NeuRx RA/4 Diaphragmatic Pacemaker in Tetraplegic Patients With Spinal Cord Injuries in Ventilator Support
Brief Title: Diaphragmatic Pacemaker in Tetraplegic Patients With Spinal Cord Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Synapse Biomedical (Industry)
Responsible Party: Principal Investigator, Miguel L. Tedde, MD, PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuRx-055110
Record Dates: First submitted 2011-06-23; First posted 2011-06-30 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Respiratory Paralysis; Diaphragmatic Paralysis; Spinal Cord Injury
MeSH Terms: conditions — Respiratory Paralysis; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NeuRx (Other)
  Interventions: Device: NeuRx RA/4 diaphragmatic pacemaker

INTERVENTIONS:
Device: NeuRx RA/4 diaphragmatic pacemaker — Patients will be implanted with 4 intramuscular electrodes, 2 in each hemi-diaphragm, using laparoscopic techniques.
  The abdominal cavity is inflated with CO2 and 4 ports are inserted: one for optics, 2 for a probe containing a temporary electrode for mapping the diaphragm and the electrode insertion tool, and a smaller one for the output wires of the electrodes of the abdominal cavity. The intra-abdominal pressure variation during the stimulation test (mapping) will be measured externally by one of the ports.
  Sites that provide the optimal response (greater region and magnitude) are noted.
  Once the optimal site for electrode placement is identified two intramuscular electrodes are deployed in each hemi-diaphragm. The guide wires will come out of the peritoneum through the port placed in the xiphoid region. An additional electrode is placed subcutaneously in the upper abdomen. The instruments and ports are then removed and the incision sites closed.

SUMMARY:
Permanent dependency of breathing apparatus due to spinal cord injury is traditionally treated with different types of mechanical ventilation. However, the electric ventilation became a possibility through their most current versions, such as diaphragmatic pacemakers.

Diaphragmatic pacemakers rhythmically stimulates the diaphragm to replace the functions of the respiratory center that doesn't works well or is inaccessible. However, this modality has the prerequisite that the phrenic nerve and diaphragm muscle are normal. The reason for the development of diaphragmatic pacemaker freeing the patient from the ventilator.

By using the mechanical energy of the diaphragm of the patient, the patient may come not need the ventilator tubing, tracheostomy, and with the help of their caregivers, the inconvenient mechanical ventilators.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Cervical spinal cord injuries patients under mechanical ventilation
* Clinically stable after spinal cord injury
* Clinical acceptable bilateral phrenic nerve function demonstrated with electromyography and neural conduction time
* Fluoroscopic visible diaphragmatic movements under stimulation
* Hemodynamically stable
* No co-morbidities that can interfere with pacemaker implantation or function
* Pregnancy negative test for women
* Patient or legal representative informed consent

Exclusion Criteria:

* Active pulmonary disease
* Active cardiovascular disease
* Active cerebral disease
* Hemodynamic instability or low oxygen levels in ambient air
* Hospitalization for infection in the last 3 months
* Significant scoliosis or chest disease
* Obesity
* Poor compliance to the protocol from the patient or the caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Volume comparison of the basal with the tidal volume obtained with the NeuRx RA/4 pacemaker in patients with diaphragmatic paralysis | One year
  The ability of the NeuRx RA / 4 to obtain clinically acceptable tidal volume during a period of 4 continuous hours will be evaluated by spirometry. Clinically acceptable volume is defined as a volume in excess of 15% above the basal metabolic requirements of the particular patient. For a male patient, the flow volume to meet the basal metabolic requirement is set at 7 ml/kg body weight, while for a female patient, it is defined in 6ml/Kg body weight.

SECONDARY OUTCOMES:
Functional rehabilitation by measure of total usage time, both day and night | One year
  Using spreadsheets to patients and caregivers, will collect information related to the use of the device, such as total usage time, the preference to use it both day and night instead of a mechanical ventilator, or to use it partial time to perform any activity or acquire independence that would otherwise be difficult with mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio B Jatene, MD, PhD, Study Director — Thoracic Surgery Department, Heart Institute (InCor) do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo; Manuel J Teixeira, MD, PhD, Study Chair — Neurosurgery Department, Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo; Miguel L Tedde, MD, PhD, Principal Investigator — Thoracic Surgery Department, Heart Institute (InCor) do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo
Locations (2):
- Brazil (2):
  - Heart Institute (InCor) Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo

REFERENCES:
- [Result] Tedde ML, Vasconcelos Filho P, Hajjar LA, de Almeida JP, Flora GF, Okumura EM, Osawa EA, Fukushima JT, Teixeira MJ, Galas FR, Jatene FB, Auler JO Jr. Diaphragmatic pacing stimulation in spinal cord injury: anesthetic and perioperative management. Clinics (Sao Paulo). 2012 Nov;67(11):1265-9. doi: 10.6061/clinics/2012(11)07. PMID 23184201
- [Result] Tedde ML, Onders RP, Teixeira MJ, Lage SG, Ballester G, Brotto MW, Okumura EM, Jatene FB. Electric ventilation: indications for and technical aspects of diaphragm pacing stimulation surgical implantation. J Bras Pneumol. 2012 Sep-Oct;38(5):566-72. doi: 10.1590/s1806-37132012000500005. English, Portuguese. PMID 23147048